CLINICAL TRIAL: NCT04406324
Title: COVID-19: Prospective Follow-up of Pulmonary Function, Sleep Disorders, Quality of Life and Post-traumatic Stress
Brief Title: COVID-19: Respiratory and Sleep Follow-up
Acronym: Co-SURVIVORS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.157
Record Dates: First submitted 2020-05-13; First posted 2020-05-28 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: COVID-19; Pulmonary function; Sleep disorders; Post-traumatic stress; Cardiac function; Sleep Apnea
MeSH Terms: conditions — COVID-19; Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 patients: Patients infected by SARS-CoV-2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention. The study consists in a prospective clinical longitudinal follow-up

SUMMARY:
The current project is a prospective, multicentric cohort study aiming at a multidisciplinary assessment (pulmonary, cardiometabolic, sleep and mental health) of the consequences of infection by SARS-CoV-2, 3 months after the diagnosis in order to better characterize these complications. 400 patients with a positive diagnosis of SARS-CoV-2 will be included in the study 3 months after their diagnosis: They will be followed at 6 months, 1 year, 3 years, and 5 years, as function of their after-effects discovered at 3 months and their evolution.

DETAILED DESCRIPTION:
Europe and in particular Italy, Spain and France are currently affected by the coronavirus 2019-nCoV pandemic, whose immediate prognosis is linked to the development of acute respiratory distress syndrome (ARDS). Beyond the long-term adverse effects on respiratory health and reduced exercise capacity, other complications will occur. These include a more rapid progression of cardiometabolic diseases, a secondary epidemic of disabling post-traumatic stress disorder, and severe sleep disorders. The current project aims at a multidisciplinary assessment of respiratory, cardiac, sleep and mental health sequelae, three months after SARS-CoV-2 diagnosis in order to better characterize these complications.

Three aspects will be targeted in this study : (i) long-term monitoring of deterioration in lung function, (ii) screening for sleep respiratory disorders (sleep apnea syndrome, obesity hypoventilation syndrome) and iii) characterization of sleep disorders and design of specialized intervention to improve sleep quality.

This study is a prospective, multicentric cohort study that aims at constituting a cohort of 400 patients who will be screened for pulmonary, cardiac, sleep, or psychological sequelae 3 months after their diagnosis. They will be then followed for 5 years. The primary outcome will be the diffusion capacity of carbon monoxide (DLCO) 3 months after the diagnosis. Other secondary outcomes will include:

* prevalence of sleep disorders and sleep disordered breathing 3 months after diagnosis and their evolution until 5 years;
* prevalence of cardiac, exercise capacity, respiratory and ventilatory muscles impairments at 3 months and their evolution until 5 years;
* characterization of homogeneous groups of patients who were infected with SARS-CoV-2 and have respiratory, cardiometabolic and/or sleep complications, 3 months after diagnosis (latent class analysis) and evaluate their evolution until 5 years
* determine the prevalence of radiological sequelae at 3 months, and their evolution until 5 years
* determine the psycho-social impact (quality of life, post-traumatic stress, anxiety, productivity at work) at 3 months and its evolution until 5 years

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged > 18 years
* With a positive diagnosis for SARS-COVID-19, confirmed by RT-PCR or with compatible symptoms
* Signed informed consent by patient
* Affiliated to a French social and health insurance system or equivalent
* For biological collection: patient eligible for sampling (weight >50kg and hemoglobin >7g/dL) and signed inform consent for collection

Exclusion Criteria:

* Pregnant or breastfeeding women
* Prisoners or patients who require protection by the law
* Patients not affiliated to a French social and health insurance system or equivalent
* Ages <18 years
* Diagnosis of infection by other pathogen than SARS-COVID-19 or no indication of infection by COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected by SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Diffusion Capacity for Carbon Monoxide (CO) 3 months after COVID diagnosis | 3 months after COVID diagnosis
  Pulmonary function 3 months after COVID diagnosis, as measured by diffusion capacity of carbon monoxide (DLCO)

SECONDARY OUTCOMES:
Prevalence of Sleep Disordered Breathing (SDB) 3 months after COVID diagnosis | 3 months after COVID diagnosis
  Prevalence of Sleep Disordered Breathing, as measured by polysomnography
Prevalence of sleep disorders 3 months after COVID diagnosis | 3 months after COVID diagnosis
  Prevalence of sleep disorders, as measured by polysomnography
Prevalence of ventilatory muscle function impairments, 3 months after COVID diagnosis | 3 months after COVID diagnosis
  Prevalence of ventilatory impairments measured by pulmonary function tests
Prevalence of cardiac impairments 3 months after COVID diagnosis | 3 months after COVID diagnosis
  Prevalence of cardiac impairments measured by cardiac echography
Follow-up of pulmonary diffusion capacity of carbon monoxide | From Baseline (3 months after COVID diagnosis) to 5 years
  Pulmonary function as measured by diffusion capacity of carbon monoxide (DLCO)
Follow-up of sleep disorders treatment compliance | From Baseline (3 months after COVID diagnosis) to 5 years
  Assessment of SDB treatments adherence will be monitored in hours/night
Follow-up of sleep disorders treatments efficacy | From Baseline (3 months after COVID diagnosis) to 5 years
  Assessment of SDB treatments efficacy will be based on the residual AHI index (Apnea Hypopnea/hour) under treatment
HLA alleles aspect of COVID clinical presentation | 3 months after COVID diagnosis
  HLA alleles will be assessed as a component of genetic immune capacity
KIR loci aspect of COVID clinical presentation | 3 months after COVID diagnosis
  KIR loci will be assessed as a different component of genetic immune capacity
metabolomic aspect of COVID clinical presentation | 3 months after COVID diagnosis
  metabolome expression in sera

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Tamisier, MD, PhD, MBA, Principal Investigator — University Hospital Grenoble Aples
Locations (4):
- France (4):
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier Henri Mondor, APHP, Créteil
  - CHU Grenoble Alpes, Grenoble
  - CHRU Nancy, Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Hui DS, Joynt GM, Wong KT, Gomersall CD, Li TS, Antonio G, Ko FW, Chan MC, Chan DP, Tong MW, Rainer TH, Ahuja AT, Cockram CS, Sung JJ. Impact of severe acute respiratory syndrome (SARS) on pulmonary function, functional capacity and quality of life in a cohort of survivors. Thorax. 2005 May;60(5):401-9. doi: 10.1136/thx.2004.030205. PMID 15860716
- [Background] Burnham EL, Hyzy RC, Paine R 3rd, Coley C 2nd, Kelly AM, Quint LE, Lynch D, Janssen WJ, Moss M, Standiford TJ. Chest CT features are associated with poorer quality of life in acute lung injury survivors. Crit Care Med. 2013 Feb;41(2):445-56. doi: 10.1097/CCM.0b013e31826a5062. PMID 23263616
- [Background] Herridge MS, Moss M, Hough CL, Hopkins RO, Rice TW, Bienvenu OJ, Azoulay E. Recovery and outcomes after the acute respiratory distress syndrome (ARDS) in patients and their family caregivers. Intensive Care Med. 2016 May;42(5):725-738. doi: 10.1007/s00134-016-4321-8. Epub 2016 Mar 30. PMID 27025938
- [Background] Luyt CE, Combes A, Becquemin MH, Beigelman-Aubry C, Hatem S, Brun AL, Zraik N, Carrat F, Grenier PA, Richard JM, Mercat A, Brochard L, Brun-Buisson C, Chastre J; REVA Study Group. Long-term outcomes of pandemic 2009 influenza A(H1N1)-associated severe ARDS. Chest. 2012 Sep;142(3):583-592. doi: 10.1378/chest.11-2196. PMID 22948576